CLINICAL TRIAL: NCT05543304
Title: Predicting Response to Systemic Therapies for Hepatocellular Carcinoma(HCC) Based on Clinical Variables and Radiomics Data With Machine Learning Methods
Brief Title: Predicting Response to Systemic Therapies for Hepatocellular Carcinoma(HCC)
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Collaborators: The First Affiliated Hospital of Zhejiang Chinese Medical University (Other); Eastern Hepatobiliary Surgery Hospital (Other); Qilu Hospital of Shandong University (Other)
Responsible Party: Principal Investigator, Gang Chen, MD, Clinical Professor, Principal Investigator, First Affiliated Hospital of Wenzhou Medical University
Other Study IDs: efficacy of systemic therapies
Record Dates: First submitted 2022-09-14; First posted 2022-09-16 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Hepatocellular Carcinoma Non-resectable; Effect of Drug
Keywords: Hepatocellular Carcinoma; systemic therapy; immunotherapy; tyrosine kinase inhibitor; treatment response; radiomics; clinical characteristics; machine learning
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with response to systemic therapies: Patients shown complete response (CR) and partial response (PR) after treatments. The clinical data and radiomics data are collected through electronic medical record system.
  Interventions: Diagnostic Test: radiological evaluation
- patients with no response to systemic therapies: Patients shown progressive disease (PD) and stable disease (SD) after treatments. The clinical data and radiomics data are collected through electronic medical record system.
  Interventions: Diagnostic Test: radiological evaluation

INTERVENTIONS:
Diagnostic Test: radiological evaluation — All patients with advanced HCC receive imaging evaluation before and after systemic treatments to assess the development of diseases.

SUMMARY:
As the most common type of primary liver cancer, hepatocellular carcinoma (HCC) has become a big challenge all over the world. Most patients are not available to curative resection when first diagnosed. There are a variety of treatment options for advanced HCC. However, due to the heterogeneity of HCC, the overall response rate (ORR) is not high for systemic therapies. Therefore, appropriate selection of patients who are suitable for individual systemic therapies is important for clinical decision-making.

DETAILED DESCRIPTION:
Although major achievements have been acquired in diagnosis and treatment, the prognosis of hepatocellular carcinoma (HCC) is still unsatisfactory. Liver resection remains the main curative treatment for HCC, but most patients are at an advanced stage when first diagnosed, leading to be not available to curative therapies. There is a variety of treatment options for advanced HCC, such as transarterial chemoembolization (TACE), hepatic artery infusion chemotherapy (HAIC), targeted therapy (sorafenib and lenvatinib), immunotherapy, and the combination of different therapies. However, due to the heterogeneity of HCC, different patients respond differently to systemic therapies. The the overall response rate (ORR) is not satisfactory and most patients can not benefit from the systemic therapies. There is an urgent need to identify patients who are likely to have positive response to systemic therapies at the beginning before treatment. Therefore ,we want to collect the clinical information of patients with advanced HCC treated with systemic therapies, including demographic data , laboratory index, histological features, radiomics data. Patients are followed-up at a interval of 1 month after treatment, and the ORR, overall survival (OS), progression-free survival (PFS) are recorded. Then the treatment response are evaluated and the relationship between the clinical data and efficacy of systemic therapies are explored by machine learning methods. Then models based on clinical features or radiomics features are developed to predict response to different systemic therapies.

ELIGIBILITY:
Inclusion Criteria:

* clinically or pathologically diagnosed HCC
* Eastern Cooperative Oncology Group performance status (ECOG-PS) 0-2
* Child-Pugh score of ≤7
* complete clinical and follow-up information
* evaluable efficacy after treatment
* age between 18-80 years old

Exclusion Criteria:

* with other malignancies
* Eastern Cooperative Oncology Group performance status (ECOG-PS) >2
* Child-Pugh score of >7
* incomplete clinical data
* lost to follow up
* unevaluable efficacy after treatment
* age <18 years old or >80 years old

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with unresectable HCC who received systemic therapies.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-12-01 (Actual); Primary Completion 2023-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective response rate | 3 months
  Tumor response are evaluated to the Modified Response Evaluation Criteria in Solid Tumors (mRECIST).

SECONDARY OUTCOMES:
Overall survival | 1 year
  Overall survival was defined as the time from treatment to death for any reason.
Progression free survival | 1 year
  Progression free survival was defined as the time from treatment to first progression or death.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Chen, MD,PhD, Principal Investigator — First Affiliated Hospital of Wenzhou Medical University
Locations (1):
- Gang Chen, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Villanueva A. Hepatocellular Carcinoma. N Engl J Med. 2019 Apr 11;380(15):1450-1462. doi: 10.1056/NEJMra1713263. No abstract available. PMID 30970190
- [Background] Llovet JM, Castet F, Heikenwalder M, Maini MK, Mazzaferro V, Pinato DJ, Pikarsky E, Zhu AX, Finn RS. Immunotherapies for hepatocellular carcinoma. Nat Rev Clin Oncol. 2022 Mar;19(3):151-172. doi: 10.1038/s41571-021-00573-2. Epub 2021 Nov 11. PMID 34764464
- [Background] Chen B, Garmire L, Calvisi DF, Chua MS, Kelley RK, Chen X. Harnessing big 'omics' data and AI for drug discovery in hepatocellular carcinoma. Nat Rev Gastroenterol Hepatol. 2020 Apr;17(4):238-251. doi: 10.1038/s41575-019-0240-9. Epub 2020 Jan 3. PMID 31900465
- [Background] Chen M, Cao J, Hu J, Topatana W, Li S, Juengpanich S, Lin J, Tong C, Shen J, Zhang B, Wu J, Pocha C, Kudo M, Amedei A, Trevisani F, Sung PS, Zaydfudim VM, Kanda T, Cai X. Clinical-Radiomic Analysis for Pretreatment Prediction of Objective Response to First Transarterial Chemoembolization in Hepatocellular Carcinoma. Liver Cancer. 2021 Feb;10(1):38-51. doi: 10.1159/000512028. Epub 2021 Jan 7. PMID 33708638
- [Background] Bruix J, Chan SL, Galle PR, Rimassa L, Sangro B. Systemic treatment of hepatocellular carcinoma: An EASL position paper. J Hepatol. 2021 Oct;75(4):960-974. doi: 10.1016/j.jhep.2021.07.004. Epub 2021 Jul 10. PMID 34256065
- [Background] Spann A, Yasodhara A, Kang J, Watt K, Wang B, Goldenberg A, Bhat M. Applying Machine Learning in Liver Disease and Transplantation: A Comprehensive Review. Hepatology. 2020 Mar;71(3):1093-1105. doi: 10.1002/hep.31103. Epub 2020 Mar 6. PMID 31907954
- [Background] Lee IC, Huang JY, Chen TC, Yen CH, Chiu NC, Hwang HE, Huang JG, Liu CA, Chau GY, Lee RC, Hung YP, Chao Y, Ho SY, Huang YH. Evolutionary Learning-Derived Clinical-Radiomic Models for Predicting Early Recurrence of Hepatocellular Carcinoma after Resection. Liver Cancer. 2021 Sep 20;10(6):572-582. doi: 10.1159/000518728. eCollection 2021 Nov. PMID 34950180